CLINICAL TRIAL: NCT04968054
Title: Comparison of Intraoperative Neurophysiological Monitoring According to the Use of Anesthetics During Total Intravenous Anesthesia in Spine Surgery Patients
Brief Title: Comparison of IONM Between Remimazolam and Propofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Dong Woo Han, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 3-2021-0189
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Ossification Posterior Longitudinal Ligament; Cervical Spondylotic Myelopathy
MeSH Terms: conditions — Ossification of Posterior Longitudinal Ligament | interventions — Propofol; remimazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol group (Active Comparator): Propofol group will be inducted and maintained total intravenous anesthesia with propofol 2% and remifentanil under Shinider and Minto target controlled infusion (TCI) model, respevtively
  Interventions: Drug: Arm I (Propofol)
- Remimazolam group (Experimental): Remimazolam group will be started total intravenous anesthesia with remiamazolam at 6 mg/kg/h at the time of anesthesia induction, and maintained at 0.5-1.5 mg/kg/h.
  Interventions: Drug: Arm II (Remimazolam)

INTERVENTIONS:
Drug: Arm I (Propofol) — Propofol group will be inducted and maintained total intravenous anesthesia with propofol 2% and remifentanil under Shinider and Minto target controlled infusion (TCI) model, respevtively.
  Arms: Propofol group
Drug: Arm II (Remimazolam) — Remimazolam group started total intravenous anesthesia with remiamazolam at 6 mg/kg/h at the time of anesthesia induction, and maintained at 0.5-1.5 mg/kg/h.
  Arms: Remimazolam group

SUMMARY:
Inhalation anesthetics significantly can delay latency and reduce amplitude of cortical MEPs and SSEPs signals compared to intravenous anesthetics by acting on not only GABA (γ-aminobutyric acid) receptors but also NMDA (N-methyl-D-aspartate) receptors, so total intravenous anesthesia (TIVA) have been more preferred for neurophysiological monitoring follow-up during surgery. However, just less than inhalation anesthetics, the decrease of amplitude and the delay of latency also occur according to the dose dependant of propofol. Moreover, it can cause various adverse effects such as delayed recovery after anesthesia or propofol infusion syndrome, consequently, combined methods with other agents or conversion to other relative anesthetics are being made. Remimazolam is a ultra-short-acting benzodiazepine, and unlike conventional benzodiazepine drugs, it is rapidly metabolized in plasma and not accumulates in the body for long periods of infusion or even with high dose administration. Recently, there have been repored that continuous infusion of 0.5-1.5 mg/kg of remimazolam has little effect on the motor evoked potential (MEPs) of cervical spine surgery patients, but this is a case report without the control group; further prospective studies are definitely needed. Therefore, in the case of using propofol or remimazolam for total intravenous anesthesia, we aim to investigate which intravenous anesthetic is more appropriate for intraoperative neurophysiological monitoring by comparing the results of the somatosensory evoked potential (SSEPs) and MEPs according to these anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who aged 20-70 years with ASA-PS 1-3, diagnosed of ossification of the posterior longitudinal ligament or cervical spondylotic myelopathy, in need of intraoperative neurophysiological monitoring

Exclusion Criteria:

* Tolerance or hypersensitivity to benzodiazepine or propofol
* Dependence or addiction to psychotropic drugs or alcohol
* Previous brain-related neurosurgery
* Inserted status of pacemaker
* Inserted status of intracranial device
* Steroids use during surgery
* Pregnant women, subjects who lack the ability to make decisions and susceptible to voluntary participation decisions

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Latency of SSEPs | At the 30 minutes after anesthetic induction (before surgical incision)
  The difference of SSEPs between the two groups (propofol vs. remimazolam) compared with baseline SSEPs

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea